CLINICAL TRIAL: NCT00822185
Title: A Single-centre, Randomised, Placebo-controlled, Double-blind, Single-dose, Dose-escalation Trial to Assess the Safety, Tolerability and Pharmacokinetics of Ascending Intravenous Doses of an Activated Recombinant FVII Analogue (NN1731) in Healthy Japanese Male Subjects
Brief Title: Safety, Tolerability and Pharmacokinetics of NN1731 in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NN1731-3604; JapicCTI-090681 (Registry Identifier: JAPIC)
Record Dates: First submitted 2009-01-13; First posted 2009-01-14 (Estimated); Results first posted 2014-09-23 (Estimated); Last update posted 2015-01-05 (Estimated); Status verified 2014-12

CONDITIONS: Congenital Bleeding Disorder; Healthy
MeSH Terms: interventions — vatreptacog alfa

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- vatreptacog alfa, 5 mcg/kg (Experimental)
  Interventions: Drug: vatreptacog alfa (activated); Drug: placebo
- vatreptacog alfa, 10 mcg/kg (Experimental)
  Interventions: Drug: vatreptacog alfa (activated); Drug: placebo
- vatreptacog alfa, 20 mcg/kg (Experimental)
  Interventions: Drug: vatreptacog alfa (activated); Drug: placebo
- vatreptacog alfa, 30 mcg/kg (Experimental)
  Interventions: Drug: vatreptacog alfa (activated); Drug: placebo

INTERVENTIONS:
Drug: vatreptacog alfa (activated) — One single dose is injected i.v. over 2 minutes to 6 subjects, 5 mcg/kg
  Arms: vatreptacog alfa, 5 mcg/kg
Drug: vatreptacog alfa (activated) — One single dose is injected i.v. over 2 minutes to 6 subjects, 10 mcg/kg
  Arms: vatreptacog alfa, 10 mcg/kg
Drug: vatreptacog alfa (activated) — One single dose is injected i.v. over 2 minutes to 6 subjects, 20 mcg/kg
  Arms: vatreptacog alfa, 20 mcg/kg
Drug: vatreptacog alfa (activated) — One single dose is injected i.v. over 2 minutes to 6 subjects, 30 mcg/kg
  Arms: vatreptacog alfa, 30 mcg/kg
Drug: placebo — Single dose is injected i.v. over 2 minutes to 2 subjects per dose level: 5 mcg/kg
  Arms: vatreptacog alfa, 5 mcg/kg
Drug: placebo — Single dose is injected i.v. over 2 minutes to 2 subjects per dose level: 10 mcg/kg
  Arms: vatreptacog alfa, 10 mcg/kg
Drug: placebo — Single dose is injected i.v. over 2 minutes to 2 subjects per dose level: 20 mcg/kg
  Arms: vatreptacog alfa, 20 mcg/kg
Drug: placebo — Single dose is injected i.v. over 2 minutes to 2 subjects per dose level: 30 mcg/kg
  Arms: vatreptacog alfa, 30 mcg/kg

SUMMARY:
This trial is conducted in Japan. The aim of this trial is to assess the safety and tolerability of activated recombinant human coagulation factor VII analogue (NN1731, vatreptacog alfa (activated)) in healthy Japanese male subjects. In addition, the pharmacokinetics of NN1731 will be examined

ELIGIBILITY:
Inclusion Criteria:

* Japanese male subjects, who are considered to be generally healthy based on assessment of medical history, physical examination and clinical laboratory data at screening, as judged by the Investigator or Sub-investigator
* Body Mass Index (BMI) between 18.0 and 27.0 kg/m^2 (inclusive)

Exclusion Criteria:

* Any clinical laboratory values deviated from the reference range at the laboratory (except for cases within physiological change) or any abnormal electrocardiogram (ECG) findings at the screening, as judged by the Investigator or Sub-investigator
* Presence or history of cancer or any clinically significant cardiac, respiratory, metabolic, renal, hepatic, gastrointestinal, endocrinological, dermatological, venereal, haematological, neurological, or psychiatric diseases or disorders
* Evidence of clinically relevant pathology or a potential thromboembolic risk as judged by the Investigator or Sub-investigator
* Presence or history of atherosclerosis, arteriosclerosis or thromboembolic events
* Any past history of migraine
* Overt bleeding, including from the gastrointestinal tract

Ages: 20 Years to 45 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 32 (Actual)
Dates: Start 2009-01; Primary Completion 2009-07 (Actual); Study Completion 2009-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Registry (GCR, 1452), Study Director — Novo Nordisk A/S
Locations (1):
- Tokyo, Japan

REFERENCES:
- See also: Clinical Trials at Novo Nordisk — http://novonordisk-trials.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This trial was conducted at a single site in Japan.
Groups:
- Vatreptacog Alfa 5 mcg/kg: A single dose of Vatreptacog alfa 5 mcg/kg bodyweight was administered intravenously
- Vatreptacog Alfa 10 mcg/kg: A single dose of Vatreptacog alfa 10 mcg/kg bodyweight was administered intravenously
- Vatreptacog Alfa 20 mcg/kg: A single dose of Vatreptacog alfa 20 mcg/kg bodyweight was administered intravenously
- Vatreptacog Alfa 30 mcg/kg: A single dose of Vatreptacog alfa 30 mcg/kg bodyweight was administered intravenously
- Placebo: A single dose of placebo was administered intravenously
Period: Overall Study
Arm/Group | Vatreptacog Alfa 5 mcg/kg | Vatreptacog Alfa 10 mcg/kg | Vatreptacog Alfa 20 mcg/kg | Vatreptacog Alfa 30 mcg/kg | Placebo
Started | 6 | 6 | 6 | 6 | 8
Completed | 6 | 6 | 6 | 6 | 8
Not Completed | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Vatreptacog Alfa 5 mcg/kg | Vatreptacog Alfa 10 mcg/kg | Vatreptacog Alfa 20 mcg/kg | Vatreptacog Alfa 30 mcg/kg | Placebo | Total
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 8 | 32
Age, Continuous [Mean (Standard Deviation); unit: years] | 28.8 (6.5) | 23.3 (3.4) | 26.5 (3.5) | 26.3 (5.1) | 26.5 (7.7) | 26.3 (5.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0 | 0 | 0 | 0
  Male | 6 | 6 | 6 | 6 | 8 | 32

OUTCOME MEASURES:

1. Primary Outcome: Safety (Physical Examination, Vital Signs, ECG, Haematology, Biochemistry, Urinalysis, Coagulation Factors, Coagulation-related Parameters, Injection Site Tolerability and Adverse Events (AE))
Description: Any safety issue was reported as AE
Time Frame: between dosing and 2-3 weeks after dosing
Population: Safety analysis set included all the randomised subjects who received at least one dose of the trial product.
Measure: Number; unit: number of events
Arm/Group | Vatreptacog Alfa 5 mcg/kg | Vatreptacog Alfa 10 mcg/kg | Vatreptacog Alfa 20 mcg/kg | Vatreptacog Alfa 30 mcg/kg | Placebo
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 8
number of events | 0 | 0 | 0 | 0 | 0

2. Primary Outcome: Subjects With Anti-Vatreptacog Alfa Antibody
Description: Post-dosing samples from subjects were evaluated for the presence of Anti-Vatreptacog alfa antibody
Time Frame: between dosing, 2-3 weeks after dosing, and 11-13 weeks after dosing
Population: Safety analysis set included all the randomised subjects who received at least one dose of the trial product.
Measure: Number; unit: participants
Arm/Group | Vatreptacog Alfa 5 mcg/kg | Vatreptacog Alfa 10 mcg/kg | Vatreptacog Alfa 20 mcg/kg | Vatreptacog Alfa 30 mcg/kg | Placebo
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 8
participants | 0 | 0 | 0 | 0 | 0

3. Secondary Outcome: Vatreptacog Alfa Clot Activity: Area Under the FVIIa Activity-time Curve From Time 0 and up Until the Last Quantifiable Activity (AUC0-t)
Description: AUC0-t was computed using the linear trapezoid rule. Plasma FVIIa clot activity at time 0 was calculated by log linear interpolation.
Time Frame: during 1-2 days after drug administration
Population: PK analysis set included all the subjects not violating the protocol in a manner that was judged to affect PK endpoint evaluation.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: (IU*h)/mL
Arm/Group | Vatreptacog Alfa 5 mcg/kg | Vatreptacog Alfa 10 mcg/kg | Vatreptacog Alfa 20 mcg/kg | Vatreptacog Alfa 30 mcg/kg
Number analyzed (Participants) | 6 | 6 | 6 | 6
(IU*h)/mL | 7.875 (10.7) | 13.845 (15.0) | 30.268 (7.5) | 46.986 (6.4)

4. Secondary Outcome: Vatreptacog Alfa Clot Activity: Area Under the FVIIa Activity-time Curve From Time 0 to 24 h (AUC0-24)
Description: Blood samples were collected at following time points: -30 min, -20 min, -10 min, 5 min, 10 min, 20 min, 30 min, 1 h, 2h, 3h, 4h, 5h, 8h, 12h and 24h to calculate area under the curve.
Time Frame: during 1-2 days after drug administration
Population: PK analysis set included all the subjects not violating the protocol in a manner that was judged to affect PK endpoint evaluation. One (1) subject did not contribute to PK evaluation.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: (IU*h)/mL
Arm/Group | Vatreptacog Alfa 5 mcg/kg | Vatreptacog Alfa 10 mcg/kg | Vatreptacog Alfa 20 mcg/kg | Vatreptacog Alfa 30 mcg/kg
Number analyzed (Participants) | 6 | 5 | 6 | 6
(IU*h)/mL | 7.970 (11.8) | 13.143 (8.1) | 30.310 (7.5) | 47.021 (6.3)

5. Secondary Outcome: Vatreptacog Alfa Clot Activity: Area Under the FVIIa Activity-time Curve From Time 0 h to Infinity (AUC 0-inf)
Description: AUC0-inf = AUC0-t + (Ct / λz), Where Ct is the last quantifiable activity and t the time of Ct.
Time Frame: during 1-2 days after drug administration
Population: as for outcome 4
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: (IU*h)/mL
Arm/Group | Vatreptacog Alfa 5 mcg/kg | Vatreptacog Alfa 10 mcg/kg | Vatreptacog Alfa 20 mcg/kg | Vatreptacog Alfa 30 mcg/kg
Number analyzed (Participants) | 6 | 5 | 6 | 6
(IU*h)/mL | 8.128 (14.7) | 13.195 (8.1) | 30.351 (7.7) | 47.060 (6.4)

6. Secondary Outcome: Vatreptacog Alfa Clot Activity: Maximum FVIIa Activity (Cmax)
Time Frame: during 1-2 days after drug administration
Population: as for outcome 3
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: IU/mL
Arm/Group | Vatreptacog Alfa 5 mcg/kg | Vatreptacog Alfa 10 mcg/kg | Vatreptacog Alfa 20 mcg/kg | Vatreptacog Alfa 30 mcg/kg
Number analyzed (Participants) | 6 | 6 | 6 | 6
IU/mL | 15.767 (10.4) | 27.569 (13.9) | 55.732 (5.9) | 86.974 (4.4)

7. Secondary Outcome: Vatreptacog Alfa Clot Activity: FVIIa Activity Measured 5 Min After Administration of NN1731 (C5min)
Time Frame: during 1-2 days after drug administration
Population: as for outcome 3
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: IU/mL
Arm/Group | Vatreptacog Alfa 5 mcg/kg | Vatreptacog Alfa 10 mcg/kg | Vatreptacog Alfa 20 mcg/kg | Vatreptacog Alfa 30 mcg/kg
Number analyzed (Participants) | 6 | 6 | 6 | 6
IU/mL | 15.767 (10.4) | 27.569 (13.9) | 55.732 (5.9) | 86.974 (4.4)

8. Secondary Outcome: Vatreptacog Alfa Clot Activity: Back Extrapolated Estimate of the Initial FVIIa Activity (C0)
Time Frame: during 1-2 days after drug administration
Population: as for outcome 3
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: IU/mL
Arm/Group | Vatreptacog Alfa 5 mcg/kg | Vatreptacog Alfa 10 mcg/kg | Vatreptacog Alfa 20 mcg/kg | Vatreptacog Alfa 30 mcg/kg
Number analyzed (Participants) | 6 | 6 | 6 | 6
IU/mL | 19.802 (8.4) | 34.497 (14.2) | 69.474 (7.3) | 106.916 (5.5)

9. Secondary Outcome: Vatreptacog Alfa Clot Activity- Terminal Slope (λz)
Time Frame: during 1-2 days after drug administration
Population: as for outcome 4
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: 1/h
Arm/Group | Vatreptacog Alfa 5 mcg/kg | Vatreptacog Alfa 10 mcg/kg | Vatreptacog Alfa 20 mcg/kg | Vatreptacog Alfa 30 mcg/kg
Number analyzed (Participants) | 6 | 5 | 6 | 6
1/h | 0.09 (59.0) | 0.14 (32.1) | 0.22 (49.9) | 0.23 (53.5)

10. Secondary Outcome: Vatreptacog Alfa Clot Activity: Terminal Half-life (t1/2)
Time Frame: during 1-2 days after drug administration
Population: PK analysis set included all the subjects not violating the protocol in a manner that was judged to affect PK endpoint evaluation. One (1) subject did not contribute to data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hours
Arm/Group | Vatreptacog Alfa 5 mcg/kg | Vatreptacog Alfa 10 mcg/kg | Vatreptacog Alfa 20 mcg/kg | Vatreptacog Alfa 30 mcg/kg
Number analyzed (Participants) | 6 | 5 | 6 | 6
hours | 7.51 (59.0) | 4.90 (32.1) | 3.14 (49.9) | 3.07 (53.5)

11. Secondary Outcome: Vatreptacog Alfa Clot Activity- Total Clearance (CL)
Time Frame: during 1-2 days after drug administration
Population: PK analysis set included all the subjects not violating the protocol in a manner that was judged to affect PK endpoint evaluation. Two (2) subjects did not contribute to data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: mL/h/kg
Arm/Group | Vatreptacog Alfa 5 mcg/kg | Vatreptacog Alfa 10 mcg/kg | Vatreptacog Alfa 20 mcg/kg | Vatreptacog Alfa 30 mcg/kg
Number analyzed (Participants) | 5 | 5 | 6 | 6
mL/h/kg | 105.14 (16.5) | 129.56 (6.3) | 110.82 (6.6) | 108.30 (6.2)

12. Secondary Outcome: Vatreptacog Alfa Clot Activity- Apparent Volume of Distribution at Steady State (Vss)
Time Frame: during 1-2 days after drug administration
Population: PK analysis set included all the subjects not violating the protocol in a manner that was judged to affect PK endpoint evaluation. Two (2) subject did not contribute to PK evaluation.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: mL/kg
Arm/Group | Vatreptacog Alfa 5 mcg/kg | Vatreptacog Alfa 10 mcg/kg | Vatreptacog Alfa 20 mcg/kg | Vatreptacog Alfa 30 mcg/kg
Number analyzed (Participants) | 5 | 5 | 6 | 6
mL/kg | 164.23 (55.0) | 131.72 (15.4) | 83.23 (18.5) | 79.67 (9.8)

13. Secondary Outcome: Vatreptacog Alfa Clot Activity- Initial Volume of Distribution (VD)
Time Frame: during 1-2 days after drug administration
Population: as for outcome 3
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: mL/kg
Arm/Group | Vatreptacog Alfa 5 mcg/kg | Vatreptacog Alfa 10 mcg/kg | Vatreptacog Alfa 20 mcg/kg | Vatreptacog Alfa 30 mcg/kg
Number analyzed (Participants) | 6 | 6 | 6 | 6
mL/kg | 43.15 (10.5) | 49.31 (15.2) | 48.41 (5.8) | 47.67 (4.9)

14. Secondary Outcome: Vatreptacog Alfa Clot Activity- Mean Residence Time (MRT)
Description: Mean residence time of the unchanged drug in the systemic circulation
Time Frame: during 1-2 days after drug administration
Population: as for outcome 4
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hours
Arm/Group | Vatreptacog Alfa 5 mcg/kg | Vatreptacog Alfa 10 mcg/kg | Vatreptacog Alfa 20 mcg/kg | Vatreptacog Alfa 30 mcg/kg
Number analyzed (Participants) | 6 | 5 | 6 | 6
hours | 1.56 (73.0) | 1.02 (14.5) | 0.75 (20.5) | 0.74 (13.0)

ADVERSE EVENTS:
Time Frame: After dosing adverse events were collected for approximately 11-13 weeks.
Description: Safety analysis set includes all subjects who received at least one dose of the investigational product or its comparator.
Arm/Group | Vatreptacog Alfa 5 mcg/kg | Vatreptacog Alfa 10 mcg/kg | Vatreptacog Alfa 20 mcg/kg | Vatreptacog Alfa 30 mcg/kg | Placebo
Serious Adverse Events (participants affected / at risk) | 0/6 | 0/6 | 0/6 | 0/6 | 0/8
Other Adverse Events (participants affected / at risk) | 0/6 | 0/6 | 0/6 | 0/6 | 0/8

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Novo Nordisk reserves the right to defer data release until specified milestones, e.g. availability of a clinical trial report. Novo Nordisk reserves the right to postpone publication and/or communication for less than 60 days to protect intellectual property. Novo Nordisk reserves the right to prior review of site-specific publications and to ask for deferment of publication of individual site results until after the primary manuscript is accepted for publication.